CLINICAL TRIAL: NCT01252706
Title: Estimation of Alcohol, Substance and Cigarettes Exposure Among Pregnant Women in the Israeli Periphery and Center, and the Contribution of Brief Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Ministry of Health, Israel (Other Government)
Responsible Party: Ariel Mani, Tel Aviv Souraski Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TASMC-10-AM-292-CTIL
Record Dates: First submitted 2010-12-01; First posted 2010-12-03 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-11

CONDITIONS: Pregnancy
Keywords: brief intervention; alcohol; nicotine; drug abuse
MeSH Terms: conditions — Substance-Related Disorders | interventions — Crisis Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: brief intervention — limit time giving information, motivation, empathy, responsibility, self control

SUMMARY:
The aims is to evaluate the rate of exposure to alcohol, psychoactive substance and nicotine among pregnant women in periphery hospital (Poria) and in the center of Tel Aviv (Ichilov) and to evaluate study Brief Intervention impact on reduction exposure, and its effect on newborn outcomes.

DETAILED DESCRIPTION:
All pregnant women who will arrive to Poria (and third of pregnant who will arrive to Ichilov) ER, high risk, and follow-up clinic will be asked for alcohol exposure, smoking and psychoactive substance usage. Relevant women will be asked to participate in a brief intervention treatment for about 30 min by expert personal, and a follow-up by phone every 3 months during pregnancy and post deliver. In addition, through all the year, questionnaires about exposure will be given to all women who will have labor (about 3000 labors), and third of 10,000 expecting in Ichilov. We expect in the second half of the year, to have those who enrolled to the BI. New-born outcome of the BI group as compared to the non-BI group will be compared, as well as rate of alcohol/substance/nicotine abstinence and reduction.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women who smoke cigarets, drink alcohol and or abuse any drugs

Exclusion Criteria:

* pregnant women who do not smoke cigarets, drink alcohol and or abuse any drugs

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10000 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-03 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
nicotine, alcohol and drug abstinence | during pregnancy until labor
  nicotine alcohol and drug abstinence will be evaluate during pregnancy until labor

SECONDARY OUTCOMES:
newborn weight of birth | at labor
  data about newborn at labor and it relation to brief intervention of mother will be deternined

CONTACTS AND LOCATIONS:
Locations (1):
- Poria Medical Center, Tiberias, Israel